CLINICAL TRIAL: NCT00934154
Title: Phase III Trial Comparing Treatment With Melphalan+Prednisolon (MP) With Melphalan+Prednisolon+Thalidomide (MPT) for Previously Untreated Elderly Patients With Multiple Myeloma
Brief Title: Melphalan+Prednisolon With or Without Thalidomide in Previously Untreated Elderly Patients With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cigdem Sahinbas YILMAZ (Industry)
Collaborators: Turkish Society of Hematology Myeloma Study Group (Unknown)
Responsible Party: Sponsor-Investigator, Cigdem Sahinbas YILMAZ, Medico Marketing Manager, Erkim Ilac A.S.
Organization: Erkim Ilac A.S. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMSG-2005-001
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-08

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; thalidomide; melphalan; prednisolone; newly diagnosed; elderly; not eligible for transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thalidomide (Experimental): MPT
  Interventions: Drug: Thalidomide; Drug: Melphalan+Prednisolone
- Control (Active Comparator): MP
  Interventions: Drug: Melphalan+Prednisolone

INTERVENTIONS:
Drug: Thalidomide — 100 mg/day continuously for 12 months
  Arms: Thalidomide
Drug: Melphalan+Prednisolone — Melphalan 2 mg, Prednisolone 16 mg

SUMMARY:
This is a multi-centre Phase III randomized controlled study of patients with multiple myeloma (MM). Eligible patients who are not candidates for transplantation will be randomized to receive eight courses of Melphalan/Prednisolone with or without Thalidomide treatment. Thalidomide will be initiated at the dose of 100 mg/day and maintained at 100 mg/day. The patients will be assessed for any responses at the end of 2nd, 4th, 6th and 8th cycles of treatment. The toxicities will be assessed at monthly intervals. Patients will be assessed for the:

1. Incidence and grade of any toxicity
2. Level of maximum disease response
3. Time to disease progression
4. Time to death

DETAILED DESCRIPTION:
This trial will include patients who are not candidates for transplantation and above the age of 55. Treatment cycles will include (MP)melphalan (9 mg /sq.m/day d1-4), prednisolone (60 mg/sq.m/d,d1-4) every six weeks for maximum 8 cycles. Patients will be randomised to (MPT) Thalidomide (1:1) 100 mg/day continuously. Cross-over to MPT is allowed if insufficient response is obtained in the MP arm. response will be evaluated every other cycle. At the end of 12 months of treatment patients will be followed until progress and death. Second line treatment is not defined.

ELIGIBILITY:
Inclusion Criteria:

* Age above 55 years old.
* Diagnosis of MM (Appendix A) and staging (Appendix B), previously untreated.
* Performance status ECOG, 0, 1, or 2 (Appendix C).
* Written informed consent to the study medications and bone marrow biopsy at diagnosis, 12 weeks and 6 months and/or off-study assessment.
* Women who are pregnant or lactating at the time of diagnosis are ineligible. All women of child-bearing potential must have a negative pregnancy test within 24hrs of commencing the thalidomide and must take adequate precautions to prevent pregnancy and should not plan on conceiving children during the treatment program:

  * Adequate precautions are defined as "at least one highly effective method i.e., IUD, hormonal (birth control pills, injections, or implants), tubal ligation, partner's vasectomy AND one additional effective method i.e., latex condom, diaphragm, cervical cap".
  * Women becoming pregnant on protocol will be removed immediately from protocol.
  * Male patients (including patients having had a vasectomy) must use barrier contraception during and for four weeks after completing the thalidomide.
* Patients remain eligible in the presence of abnormal renal function and/or liver function at time of enrollment.
* Absence of severe dementia, able to take medication at home.
* Absence of systemic disorders (gastrointestinal, pulmonary, cardiac and neurological).

Exclusion Criteria:

* Asymptomatic myeloma or solitary plasmacytoma of bone or extramedullary plasmacytoma (without evidence of myeloma).
* Previous or concurrent active malignancies, except surgically removed basal cell carcinoma of the skin or other in situ carcinomas.
* Previous treatment for myeloma, except minimal local radiotherapy to relieve bone pain.
* Other illnesses which would preclude chemotherapy administration or patient compliance.
* Any other serious medical or psychiatric illness which would prevent informed consent.
* Peripheral neuropathy > NCI criteria grade 2.
* Pregnant or lactating women and patients of childbearing age who refuse to use contraception.
* History of hypersensitivity to thalidomide or any component of the medications.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2006-03; Primary Completion 2009-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
response rate | 12 months

SECONDARY OUTCOMES:
time to relapse | 18 months
overall survival | unlimited

CONTACTS AND LOCATIONS:
Overall Officials: Meral Beksac, Prof.Dr., Principal Investigator — Ankara University; Rauf Haznedar, Prof.Dr., Principal Investigator — Gazi University
Locations (9):
- Turkey (Türkiye) (9):
  - Baskent University School of Medicine Education and Research Hospital, Hematology Department, Adana
  - Ankara Numune Education and Research Hospital,Hematology Department, Ankara
  - Ankara University School of Medicine, Hematology Department, Ankara
  - Gazi University School of Medicine, Hematology Department, Ankara
  - Hacettepe University School of Medicine, Hematology Department, Ankara
  - Akdeniz University School of Medicine , Hematology Department, Antalya
  - Uludag University School of Medicine, Hematology Department, Bursa
  - Osmangazi University School of Medicine , Hematology Department, Eskişehir
  - Marmara University School of Medicine, Hematology Department, Istanbul

REFERENCES:
- [Derived] Beksac M, Haznedar R, Firatli-Tuglular T, Ozdogu H, Aydogdu I, Konuk N, Sucak G, Kaygusuz I, Karakus S, Kaya E, Ali R, Gulbas Z, Ozet G, Goker H, Undar L. Addition of thalidomide to oral melphalan/prednisone in patients with multiple myeloma not eligible for transplantation: results of a randomized trial from the Turkish Myeloma Study Group. Eur J Haematol. 2011 Jan;86(1):16-22. doi: 10.1111/j.1600-0609.2010.01524.x. Epub 2010 Nov 22. PMID 20942865